CLINICAL TRIAL: NCT07275450
Title: Safety and Efficacy of Regional Anesthesia for Awake Tympanoplasty Surgery: A Randomized Controlled Trial
Brief Title: Comparative Study Between Ultrasound Guided Regional Anesthesia for Awake Tympanoplasty Surgery vs General Anesthesia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Dina Abdelhameed Elsadek Salem, Associate professor of anesthesia, Zagazig University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1841
Record Dates: First submitted 2025-11-25; First posted 2025-12-10 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-11

CONDITIONS: Ultrasound Guided Nerve Block; Anesthesia , Analgesia
Keywords: Ultrasound guided regional anesthesia; General anesthesia; Awake tympanoplasty
MeSH Terms: conditions — Agnosia | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: To evaluate ultrasound-guided regional anesthesia versus general anesthesia in patients undergoing tympanoplasty
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ultrasound-guided regional anesthesia group (Active Comparator): patients will receive regional anesthesia using ultrasound guidance. Target nerves (e.g., great auricular nerve, auriculotemporal nerve and lesser occipital nerve) will be identified and anesthetized under real-time ultrasound visualization to ensure accurate needle placement and local anesthetic spread.
  Interventions: Procedure: Ultrasound-guided regional anesthesia group
- Control group (Sham Comparator): patients will receive general anesthesia
  Interventions: Other: Control group

INTERVENTIONS:
Procedure: Ultrasound-guided regional anesthesia group — patients will receive regional anesthesia using ultrasound guidance. Target nerves (e.g., great auricular nerve, auriculotemporal nerve and lesser occipital nerve) will be identified and anesthetized under real-time ultrasound visualization to ensure accurate needle placement and local anesthetic spread.
  Arms: Ultrasound-guided regional anesthesia group
Other: Control group — patients will receive general anesthesia.
  Arms: Control group

SUMMARY:
The aim of this study to evaluate efficacy of ultrasound guided regional anesthesia in performing awake tympanoplasty surgery versus traditional general anesthesia

DETAILED DESCRIPTION:
* To evaluate ultrasound-guided regional anesthesia versus general anesthesia in patients undergoing tympanoplasty as regards:
* To assess the time of discharge from post anesthesia care unit
* To assess intraoperative hemodynamic parameters, quality of the surgical field and the block success rate (number of patients converted to general anesthesia).
* To assess postoperative parameters: Numerical Rating Scale , time to first request of analgesia, postoperative opioid consumption, patient and surgeon satisfaction in both groups.
* To assess the incidence of block-related complications (such as nerve injury, hematoma, inadequate block, or local anesthetic toxicity) or surgery related complications as nausea and vomiting

ELIGIBILITY:
Inclusion Criteria:

1. Patients acceptance
2. Age: 21-65 years old
3. Sex: both sex (males or females).
4. Physical status: American Society Anesthesiologist (ASA) І and II.
5. Patients will be scheduled for elective unilateral tympanoplasty.

Exclusion Criteria:

1. Contraindication of regional anesthesia: Coagulopathy or use of anticoagulant therapy -local infection at the site of injection- known allergy to local anesthetics (bupivacaine).
2. Neurological disorders affecting sensation in the head and neck.
3. Psychiatric illness, severe anxiety, or inability to cooperate during awake surgery.
4. History of previous neck or parotid surgery affecting nerve anatomy.
5. BMI > 35 (if it may interfere with ultrasound visualization or landmark identification).
6. Pregnancy.
7. Advanced cardiovascular, respiratory, hepatic and renal diseases

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 128 (Estimated)
Dates: Start 2025-12-10 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
The time of discharge from Post Anesthesia Care Unit (PACU) | 2 hours postoperative
  The time from arrival to the Post Anesthesia Care Unit (PACU) to the time to discharge to the ward according to modified aldrete score

SECONDARY OUTCOMES:
Intraoperative mean arterial blood pressure | 0 minute (basal) and every 5 minutes up to 2 hours
  Intraoperative changes in mean arterial blood pressure (mmHg)
Pain intensity by using Numerical Rating Scale (NRS) | Post Anesthesia Care Unit (0 hour) , 2 hours, 4 hours, 8 hours, 12 hours and 24 hours
  It is a scale from 0 to 10, where 0=no pain and 10= worst pain
Block success rate | 15-20 minutes (from finishing block till start surgery)
  The number of patients converted to general anesthesia
Quality of surgical field | duration of surgery (intraoperative)
  quality of surgical field by Modena Bleeding Score (MBS) is a validated categorical scale designed to measure the quality of the surgical field in relation to bleeding during endoscopic surgery. It features five grades (1= no bleeding, 2= bleeding easily controlled by suction, 3= bleeding that slows surgical procedure, 4= most maneuvers are dedicated to bleeding control and 5= bleeding is so sever that only procedures aimed at controlling bleeding)
Time to first request of analgesia | 24 hours
  Time to first request of analgesia (pethidine)
Total postoperative analgesic consumption | 24 hours
  total postoperative pethidine consumption
Patient satisfaction by Likert score | 24 hours
  patient satisfaction by Likert score: The patients will be asked to rate the overall degree of satisfaction of the analgesia by using a 5-points Likert-like verbal scale (1 = very dissatisfied analgesia, 2 = dissatisfied analgesia, and 3 = neutral, 4=satisfied analgesia, and 5=very satisfied analgesia)
Surgeon satisfaction | duration of surgery (intraoperative)
  Surgeon satisfaction by asking the surgeon to rate satisfaction at the end of surgery (4 =excellent, 3=good, 2=fair, 1=poor, 0=extremely poor)
The incidence of block-related complications or surgery related complications | 24 hours
  To assess the incidence of block-related complications, such as nerve injury, hematoma, inadequate block, or local anesthetic toxicity or surgery related complications (e.g. nausea and vomiting)
Intraoperative heart rate ( beat per minute) | before starting anesthesia 0 minute (basal )and every 5 minutes up to 2 hours
  measure intraoperative changes in heart rate

CONTACTS AND LOCATIONS:
Locations (1):
- faculty of human medicine, Zagazig university hospitals, Zagazig, Egypt

IPD SHARING:
Plan to Share IPD: No